CLINICAL TRIAL: NCT06246084
Title: INTENT Pilot Study - Enhancing Adherence Intentions to Endocrine Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Ann H. Partridge, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-607
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Breast Cancer Female; Breast Carcinoma
Keywords: Breast Cancer; Breast Cancer Female; Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Endocrine Therapy Education Intervention (Experimental): Participants will complete:
  * Baseline visit.
  * Educational video once a week for 6 weeks.
  * 6-week survey.
  * 3-month survey.
  Interventions: Behavioral: Endocrine Therapy Education Program
- Group B: Wait-List Control Group (No Intervention): Participants will complete:
  * Baseline visit.
  * 6-week survey.
  * 3-month survey.
  * Access to intervention educational videos.
  * 2-week post video survey.

INTERVENTIONS:
Behavioral: Endocrine Therapy Education Program — Brief, video-based intervention program to improve endocrine therapy adherence and experiences and to provide detailed education to participants. The intervention is distributed and assessed via the MyEmma platform, a HIPAA-compliant, online communications platform.
  Arms: Group A: Endocrine Therapy Education Intervention

SUMMARY:
This research is being done to pilot an intervention which aims to improve participants' experiences on Endocrine Therapy.

The name of the intervention used in this research study is:

Endocrine Therapy Education Program (a brief, video-based intervention)

DETAILED DESCRIPTION:
This research study is a randomized pilot study to determine whether a brief-video based intervention program can improve experiences of Endocrine Therapy (ET). Participants will be randomized into one of two groups: Group A: Endocrine Therapy Education Intervention vs. Group B Wait-list Control Group. Randomization means a participant is placed into a study group by chance.

The research study procedures include screening for eligibility, in-clinic visits, and survey questionnaires.

Participation in this research study is expected to last 3 months.

It is expected that about 60 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Biologically female
* About to begin or just started (within four weeks of starting) an oral form of ET (either tamoxifen or AI)
* 18 years of age or older
* English fluency for reading and writing.
* Computer literacy (ability to watch videos and fill out questionnaires online)

Exclusion Criteria:

* Adults unable to consent
* Individuals with metastatic cancer
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 76 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Engagement Rate of Intervention | 6 weeks
  Adequate engagement of the intervention is defined as a click-to-open rate of 60% or over for the intervention group.
Intervention Satisfaction Questionnaire Mean Score Group A | At 6 weeks
  Responses will be analyzed to determine a mean score for each item for the intervention group. The Intervention Satisfaction Questionnaire includes 9 items rated on a 1 to 10 scale.
Intervention Satisfaction Questionnaire Mean Score Group B | At 14 weeks
  Responses will be analyzed to determine a mean score for each item for the control group (following the release of the intervention educational videos). The Intervention Satisfaction Questionnaire includes 9 items rated on a 1 to 10 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Partridge, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu
URL: https://www.dana-farber.org/research/innovations